CLINICAL TRIAL: NCT05352035
Title: A Multiomics Study of Tumor Evolution Characteristics and Prognostic Model in Early-stage Non-small Cell Lung Cancer
Brief Title: Multiomics Tumor Evolution Model of NSCLC
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Research Unit of Intelligence Diagnosis and treatment of early-stage non-small cell lung cancer, Chinese Academy of Medical Sciences (Unknown)
Responsible Party: Principal Investigator, Jun Wang, Member of the Chinese Academy of Engineering, Peking University People's Hospital
Other Study IDs: 2021-I2M-5-002
Record Dates: First submitted 2022-04-23; First posted 2022-04-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Multiomics analysis; Tumor evolution; Tumor immune microenvironment; Circulating tumor DNA; Radiomics; Prognostic model
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort: This cohort will enroll a total of 300 patients prospectively

SUMMARY:
The purpose of this study is to determine the evolutionary mechanism of early-stage non-small cell lung cancer and establish an accurate prognostic model and a recurrence monitoring system by multiomics analysis, which can be helpful for the individual and whole management of lung cancer patients and improve the overall prognosis.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death globally. Non-small cell lung cancer (NSCLC) accounts for 85% of lung cancer and surgery is still the main treatment strategy. This study will determine the evolutionary mechanism of early-stage non-small cell lung cancer and establish an accurate prognostic model and a recurrence monitoring system by multiomics analysis, which can be helpful for the individual and whole management of lung cancer patients and improve the overall prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Early-stage NSCLC patients underwent radical surgical resection;
3. Sufficient tumor tissue and blood sample for study use;
4. Available clinical-pathologic data, imaging data and follow-up date;
5. Written informed consent.

Exclusion Criteria:

1. History of other malignant tumors;
2. Evidence of distant metastasis before surgery;
3. Insufficient tumor tissue or blood sample for study use;
4. Clinical-pathologic data, imaging data or follow-up date is not available;
5. Other judgments by the Investigator that the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the eligibility criteria will be included consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Through study completion, an average of 2 years
  Time from randomization to disease recurrence or death from any cause.
Overall survival (OS) | Through study completion, an average of 2 years
  Time from randomization to death from any cause.

SECONDARY OUTCOMES:
Relationship between translational biomarkers and clinical outcome | Through study completion, an average of 2 years
  To evaluate if the translational biomarkers can be prediction tools for the clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided